CLINICAL TRIAL: NCT02709135
Title: Can Pre-Hospital Use of the HEART Score and Abbott i-STAT® Point-of-Care Troponin Predict Major Adverse Cardiovascular Events: the PARA-HEART Pilot Implementation
Brief Title: PARA-HEART Pilot Implementation
Acronym: PARA-HEART
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00036229
Record Dates: First submitted 2016-03-03; First posted 2016-03-15 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2018-09

CONDITIONS: Acute Coronary Syndrome; Chest Pain
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-hospital HEART Score: All subjects included in this quality surveillance study will have had a HEART score, including POC troponin calculated by paramedics prior to arrival at the emergency department.

SUMMARY:
Approximately 8-10 million patients complaining of chest pain present to an Emergency Department (ED) annually in the United States. These patients are a challenge to healthcare providers, who are tasked with determining whether these symptoms are due to an acute coronary syndrome (ACS) or a non-ACS cause.In an effort to improve the quality and value of care for patients with acute chest pain, our group recently validated a risk stratification pathway, the HEART Pathway, which is designed to focus cardiac testing and admissions on higher-risk patients, who are more likely to benefit from testing.While the HEART score has been well validated in the ED setting, it has yet to be implemented in a prehospital setting. Paramedics are often the first providers to evaluate and begin treating patients with symptoms concerning for ACS. Current pre-hospital risk stratification is largely based on a combination of ECG results and paramedic gestalt. Since ECGs without signs of a STEMI (ST-segment elevation myocardial infarction) are poor predictors of ACS, paramedics often have difficulty distinguishing high-risk patients from low-risk patients.Thus, multidisciplinary leaders within Emergency Medicine, Cardiology, and Prehospital Medicine have agreed that a limited/pilot evaluation of the HEART Score with Abbott's i-STAT® point-of-care (POC) troponin testing in the prehospital setting is needed. To establish the feasibility and accuracy of HEART score and POC testing in the prehospital setting the investigators propose a quality surveillance study of a limited implementation of the HEART score with POC troponin testing.

DETAILED DESCRIPTION:
Approximately 8-10 million patients complaining of chest pain present to an Emergency Department (ED) annually in the United States. These patients are a challenge to healthcare providers, who are tasked with determining whether these symptoms are due to an acute coronary syndrome (ACS) or a non-ACS cause. Missing the diagnosis of ACS is associated with high rates of morbidity, mortality, and malpractice claims. Therefore, to avoid missing the diagnosis of ACS, patients with chest pain typically undergo extensive evaluations at an estimated cost of $10-13 billion annually. However, less than 10% of these patients are ultimately diagnosed with ACS. As the US healthcare system shifts towards a value-based model, it is clear that the current care patterns for acute chest pain, which fail to focus health system resources, such as hospitalization and cardiac testing, on patients most likely to benefit, are not sustainable.

In an effort to improve the quality and value of care for patients with acute chest pain, our group recently validated a risk stratification pathway, the HEART Pathway, which is designed to focus cardiac testing and admissions on higher-risk patients, who are more likely to benefit from testing. The HEART Pathway, which utilizes an easy to use clinical decision aid (the HEART score) and serial troponin measurement, has been shown to significantly reduce objective cardiac testing (stress testing and coronary angiography), shorten hospital length of stay, and increase the early discharge rate from the Emergency Department among patients with acute chest pain. These important efficiency gains occur without missing ACS and without increasing return visits to the ED or downstream admissions to the hospital over a 30 day period.

While the HEART score has been well validated in the ED setting, it has yet to be implemented in a prehospital setting. Paramedics are often the first providers to evaluate and begin treating patients with symptoms concerning for ACS. Current pre-hospital risk stratification is largely based on a combination of ECG results and paramedic gestalt. Since ECGs without signs of a STEMI are poor predictors of ACS, paramedics often have difficulty distinguishing high-risk patients from low-risk patients. Therefore, integrating objective risk stratification tools, such as the HEART score and point-of-care troponin testing, into Emergency Medical Services (EMS) triage and destination plans represents an opportunity to improve care. Furthermore, expanding use of the HEART score to paramedics in the pre-hospital setting is a natural extension of our prior work, especially given the growing sophistication of mobile integrated healthcare ("community paramedicine") over the last decade. Thus, multidisciplinary leaders within Emergency Medicine, Cardiology, and Prehospital Medicine have agreed that a limited/pilot evaluation of the HEART Score with Abbott's i-STAT® point-of-care (POC) troponin testing in the prehospital setting is needed.

The investigators anticipate that a standardized approach to paramedic risk stratification using the HEART score with Abbott's i-STAT® POC troponin testing will be feasible and achieve high accuracy for the detection of ACS. Ultimately the investigators believe this planned implementation will improve the quality and value of chest pain care. Placing these tools in the hands of our first responders will identify patients with ACS earlier and speed the delivery of potentially life-saving care. For example, EMS triage and destination plans (chest pain treatment and transportation triage and destination plans) could be amended so that patients with positive POC troponins or high HEART scores could be transported directly to a hospital with cardiac catheterization capabilities, avoiding delays and costs associated with inter-facility transfers. However, before EMS triage and destination plans can fully incorporate the HEART score and POC troponin testing, first the feasibility of such an implementation must be established by collecting quality surveillance data.

To establish the feasibility and accuracy of HEART score and POC testing in the prehospital setting the investigators propose a quality surveillance study of a limited implementation of the HEART score with POC troponin testing. This pilot will include paramedics from three demographically distinct counties (Forsyth, Surry, and Stokes counties) in North Carolina, who will begin using the HEART score and i-STAT POC Troponin as part of their risk assessment for patients with acute chest pain. However, EMS triage and transportation plans will not be altered based on the HEART score assessment until feasibility and accuracy have been established. To ensure the feasibility and accuracy of paramedic chest pain risk assessment the investigators will be performing surveillance of electronic health records (EHR) and contacting patients by phone (which is a common practice in EMS quality assurance). Quality surveillance participants (n=500) will be identified retrospectively and quality assurance data will be collected electronically using EHR (EMS records, and Wake Forest Baptist Health health records) and via telephone follow-up calls (which are customary in EMS quality assurance projects).

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 21 years
* Non-traumatic chest discomfort or other symptoms consistent with possible
* Patient being transported to Wake Forest Baptist Health ED for further care

Exclusion Criteria:

* ST-segment elevation in contiguous leads on any electrocardiogram
* Inter-facility transfers
* Short Pre-hospital times: anticipated scene + transportation time less than 5 mins
* Unstable vitals signs
* Known terminal diagnosis with life expectancy less than 1 year
* Concomitant non-cardiac medical, surgical, or psychiatric emergency

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with symptoms concerning for acute coronary syndrome who are being transported to the Wake Forest Baptist Medical Center Emergency Department by paramedics trained to complete a HEART Score and POC troponin assessment will be eligible for inclusion in this quality surveillance study.
Sampling Method: Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) at 30 days | 30 Days
  The primary outcome is MACE at 30 days. MACE is a composite outcome of cardiac death, acute myocardial infarction, and coronary revascularization.

SECONDARY OUTCOMES:
Rate of objective cardiac testing | 30 Days
  Objective cardiac testing will be defined by any stress testing modality, coronary computed tomography (CT) angiography, or invasive coronary angiography.
Length of Stay | 30 Days
  Length of stay (LOS) will be the time from ED arrival to hospital discharge for all patients, whether admitted or not.
Rate of hospitalization at index | 30 Days
  Index visit hospitalization will be defined as an inpatient or observation admission (including Observation Unit evaluations with stress testing or cardiac imaging).
Rate of cardiac related hospital admissions and ED visits during follow-up | 30 Days
  Hospital admissions and ED visits occurring during the 30 day follow up period will be categorized as cardiac-related if a cardiac procedure is performed, the primary reason for admission/visit is chest pain, possible ACS, or a discharge diagnosis relates to chest pain, myocardial infarction (MI), acute coronary syndrome, heart failure, dysrhythmias, pericardial disease, or other cardiac disease. Cardiac procedures include cardiac imaging / stress testing (excluding resting echo), coronary revascularization, and pacemaker or defibrillator insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Mahler, MD, MS, Principal Investigator — Associate Professor
Locations (1):
- Wake Forest School Of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] McCaig LF, Nawar EW. National Hospital Ambulatory Medical Care Survey: 2004 emergency department summary. Adv Data. 2006 Jun 23;(372):1-29. PMID 16841785
- [Background] Owens PL, Barrett ML, Gibson TB, Andrews RM, Weinick RM, Mutter RL. Emergency department care in the United States: a profile of national data sources. Ann Emerg Med. 2010 Aug;56(2):150-65. doi: 10.1016/j.annemergmed.2009.11.022. Epub 2010 Jan 15. PMID 20074834
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Pines JM, Isserman JA, Szyld D, Dean AJ, McCusker CM, Hollander JE. The effect of physician risk tolerance and the presence of an observation unit on decision making for ED patients with chest pain. Am J Emerg Med. 2010 Sep;28(7):771-9. doi: 10.1016/j.ajem.2009.03.019. Epub 2010 Feb 25. PMID 20837253
- [Background] Fleischmann KE, Goldman L, Johnson PA, Krasuski RA, Bohan JS, Hartley LH, Lee TH. Critical pathways for patients with acute chest pain at low risk. J Thromb Thrombolysis. 2002 Apr;13(2):89-96. doi: 10.1023/a:1016246814235. PMID 12101386
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Heller GV, Stowers SA, Hendel RC, Herman SD, Daher E, Ahlberg AW, Baron JM, Mendes de Leon CF, Rizzo JA, Wackers FJ. Clinical value of acute rest technetium-99m tetrofosmin tomographic myocardial perfusion imaging in patients with acute chest pain and nondiagnostic electrocardiograms. J Am Coll Cardiol. 1998 Apr;31(5):1011-7. doi: 10.1016/s0735-1097(98)00057-6. PMID 9562001
- [Background] Sprivulis PC, Da Silva JA, Jacobs IG, Frazer AR, Jelinek GA. The association between hospital overcrowding and mortality among patients admitted via Western Australian emergency departments. Med J Aust. 2006 Mar 6;184(5):208-12. doi: 10.5694/j.1326-5377.2006.tb00416.x. PMID 16515429
- [Background] Miro O, Antonio MT, Jimenez S, De Dios A, Sanchez M, Borras A, Milla J. Decreased health care quality associated with emergency department overcrowding. Eur J Emerg Med. 1999 Jun;6(2):105-7. doi: 10.1097/00063110-199906000-00003. PMID 10461551
- [Background] Six AJ, Backus BE, Kelder JC. Chest pain in the emergency room: value of the HEART score. Neth Heart J. 2008 Jun;16(6):191-6. doi: 10.1007/BF03086144. PMID 18665203
- [Background] Backus BE, Six AJ, Kelder JC, Mast TP, van den Akker F, Mast EG, Monnink SH, van Tooren RM, Doevendans PA. Chest pain in the emergency room: a multicenter validation of the HEART Score. Crit Pathw Cardiol. 2010 Sep;9(3):164-9. doi: 10.1097/HPC.0b013e3181ec36d8. PMID 20802272
- [Background] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250
- [Background] Mahler SA, Miller CD, Hollander JE, Nagurney JT, Birkhahn R, Singer AJ, Shapiro NI, Glynn T, Nowak R, Safdar B, Peberdy M, Counselman FL, Chandra A, Kosowsky J, Neuenschwander J, Schrock JW, Plantholt S, Diercks DB, Peacock WF. Identifying patients for early discharge: performance of decision rules among patients with acute chest pain. Int J Cardiol. 2013 Sep 30;168(2):795-802. doi: 10.1016/j.ijcard.2012.10.010. Epub 2012 Oct 30. PMID 23117012
- [Background] Mahler SA, Hiestand BC, Goff DC Jr, Hoekstra JW, Miller CD. Can the HEART score safely reduce stress testing and cardiac imaging in patients at low risk for major adverse cardiac events? Crit Pathw Cardiol. 2011 Sep;10(3):128-33. doi: 10.1097/HPC.0b013e3182315a85. PMID 21989033
- [Background] Mahler SA, Riley RF, Hiestand BC, Russell GB, Hoekstra JW, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Elliott SB, Herrington DM, Burke GL, Miller CD. The HEART Pathway randomized trial: identifying emergency department patients with acute chest pain for early discharge. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2):195-203. doi: 10.1161/CIRCOUTCOMES.114.001384. Epub 2015 Mar 3. PMID 25737484
- [Background] Hollander JE, Blomkalns AL, Brogan GX, Diercks DB, Field JM, Garvey JL, Gibler WB, Henry TD, Hoekstra JW, Holroyd BR, Hong Y, Kirk JD, O'Neil BJ, Jackson RE; Multidisciplinary Standardized Reporting Criteria Task Force. Standardized reporting guidelines for studies evaluating risk stratification of ED patients with potential acute coronary syndromes. Acad Emerg Med. 2004 Dec;11(12):1331-40. doi: 10.1197/j.aem.2004.08.033. No abstract available. PMID 15576525
- [Background] Venturini JM, Stake CE, Cichon ME. Prehospital point-of-care testing for troponin: are the results reliable? Prehosp Emerg Care. 2013 Jan-Mar;17(1):88-91. doi: 10.3109/10903127.2012.717166. Epub 2012 Sep 6. PMID 22954226
- [Background] Stengaard C, Sorensen JT, Ladefoged SA, Christensen EF, Lassen JF, Botker HE, Terkelsen CJ, Thygesen K. Quantitative point-of-care troponin T measurement for diagnosis and prognosis in patients with a suspected acute myocardial infarction. Am J Cardiol. 2013 Nov 1;112(9):1361-6. doi: 10.1016/j.amjcard.2013.06.026. Epub 2013 Aug 14. PMID 23953697
- [Background] Sorensen JT, Terkelsen CJ, Steengaard C, Lassen JF, Trautner S, Christensen EF, Nielsen TT, Botker HE, Andersen HR, Thygesen K. Prehospital troponin T testing in the diagnosis and triage of patients with suspected acute myocardial infarction. Am J Cardiol. 2011 May 15;107(10):1436-40. doi: 10.1016/j.amjcard.2011.01.014. Epub 2011 Mar 15. PMID 21414596
- [Background] Kline JA, Mitchell AM, Runyon MS, Jones AE, Webb WB. Electronic medical record review as a surrogate to telephone follow-up to establish outcome for diagnostic research studies in the emergency department. Acad Emerg Med. 2005 Nov;12(11):1127-33. doi: 10.1197/j.aem.2005.04.012. Epub 2005 Sep 15. PMID 16166598
- [Background] Havas S. The ACCORD Trial and control of blood glucose level in type 2 diabetes mellitus: time to challenge conventional wisdom. Arch Intern Med. 2009 Jan 26;169(2):150-4. doi: 10.1001/archinternmed.2008.518. No abstract available. PMID 19171811
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Derived] Stopyra JP, Snavely AC, Smith LM, Harris RD, Nelson RD, Winslow JE, Alson RL, Pomper GJ, Riley RF, Ashburn NP, Hendley NW, Gaddy J, Woodrum T, Fornage L, Conner D, Alvarez M, Pflum A, Koehler LE, Miller CD, Mahler SA. Prehospital use of a modified HEART Pathway and point-of-care troponin to predict cardiovascular events. PLoS One. 2020 Oct 7;15(10):e0239460. doi: 10.1371/journal.pone.0239460. eCollection 2020. PMID 33027260